CLINICAL TRIAL: NCT06443008
Title: Objective To Investigate the Effect of Myoelectric Biofeedback Therapy Combined With Comprehensive Rehabilitation Training on Upper Extremity Motor Function in Elderly Patients With Hemiplegia With Cerebral Infarction
Brief Title: Effects of Myoelectric Biofeedback on Upper Limb Function in Post-stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-099
Record Dates: First submitted 2024-05-28; First posted 2024-06-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Biofeedback; Rehabilitation; Cerebral Infarction
Keywords: Rehabilitation treatment; upper extremity motor function; emg biofeedback; cerebral infarction
MeSH Terms: conditions — Cerebral Infarction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Comprehensive rehabilitation treatment in control group
- Observation Group (Experimental): The observation group carried out myoelectric biofeedback therapy on the basis of the control group
  Interventions: Device: Observation Group

INTERVENTIONS:
Device: Observation Group — On the basis of myoelectric biofeedback treatment in the control group, the control group was trained alternately in each muscle group (triangle muscle, triceps brachii muscle group and forearm extensor muscle group). For example,After disinfection of the triangular, triceps and extensor muscles of the patient, the feedback electrode was attached to the area. The stimulation frequency was set at 50 Hz and the stimulation pulse width was set at 200 μs.During treatment, the patient is instructed to listen carefully to the device's password, drive the affected limb according to the specific password, and then perform tension and relaxation training.For each muscle group, the training time of each muscle group is about 0.5 h, 1 / d.In the later stage of treatment, the training intensity can be increased appropriately, so that the patient can carry out weight lifting during the feedback treatment, and listen to the password issued by the device to carry out muscle strength exercise.
  Arms: Observation Group

SUMMARY:
The purpose of this clinical trial is to investigate the effect of myoelectric biofeedback therapy on upper limb function in elderly patients with cerebral infarction, and to analyze the adjustment of stroke condition and quality of life.The main questions it aims to answer are:

1. Does myoelectric biofeedback therapy promote the restoration of upper limb function in elderly patients with cerebral infarction?
2. What medical problems do participants have with myoelectric biofeedback therapy?

DETAILED DESCRIPTION:
We divided the participants into control group and observation group using simple random method.We will number the numbers according to the order of inclusion: then from any row in the random number table as a starting point, we will get a random number sequentially from its series of numbers, paired with the included case number, and list the random distribution table.The control group was represented by odd numbers of random tables and even numbers by observation groups.The probability of being included in the control group and the observation group were 50% respectively.The control group underwent comprehensive rehabilitation training, and the observation group conducted myoelectric biofeedback treatment on the basis of the control group.

Control group treatment plan

1. After stroke, medical staff should adjust the position of the patient every 2 hours, so that the patient's position is adjusted between the healthy side position and other positions, and provide the patient with soft pillow limit.
2. Passive training, in the initial physical disability of the patient after treatment by the rehabilitation therapist to provide passive training for the patient, specifically by the rehabilitation therapist on the affected side joint.
3. Anti-spasmodic activities, through the patient's activity training to avoid spastic symptoms, help the patient to change the posture to a healthy side position before the training begins.
4. At the beginning of the training, the rehabilitation therapist places both hands under the patient's shoulder blades, so that the patient's shoulders and shoulder blades are stretched forward to help the patient stay seated.In addition, the patient is provided with Bobas handshake training to maintain the trunk forward tilt position during the training process, maintaining the center of gravity below, helping the patient to stay seated for a long time for balance training.
5. Active training, the rehabilitation therapist instructs the patient to put the hand on the prepared cushion in advance, and then let the patient use both upper limbs to stretch the fixed elastic band to implement impedance training.After the above activities can be completed, you can try to implement refined operations, including threading and other activities that require high hand activities.After the patient's upper limb function has been restored, he or she can conduct autonomous life ability training under the guidance of a rehabilitation therapist, including basic activities such as getting up and washing.The pre-active training training time is maintained at about 0.5 h, and the maximum number of training times in one day is 3 times, and the intensity of training can be increased appropriately after the patient's physical condition has recovered.

Observation group treatment plan

The observation group carried out myoelectric biofeedback therapy on the basis of the control group:

After disinfection of the triangular, triceps and extensor muscles of the patient, the feedback electrode was attached to the area. The stimulation frequency was set at 50 Hz and the stimulation pulse width was set at 200 μs.During treatment, the patient is instructed to listen carefully to the device's password, drive the affected limb according to the specific password, and then perform tension and relaxation training.For each muscle group, the training time of each muscle group is about 0.5 h, 1 / d.In the later stage of treatment, the training intensity can be increased appropriately, so that the patient can carry out weight lifting during the feedback treatment, and listen to the password issued by the device to carry out muscle strength exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Subject volunteered to participate in the experiment and signed informed consent
2. Age ≥ 65 years old, no gender limit;
3. Diagnosis of stroke patients;
4. No other major cardiovascular diseases

Exclusion Criteria:

1. Subject's poor compliance
2. Subjects with skin allergies
3. Those who do not meet the criteria for diagnosis and inclusion;
4. People with severe consciousness disorders, severe dementia, speech disorders, etc. who are unable to communicate and describe the disease;
5. can not cooperate as required, poor compliance;
6. participants in other clinical trials;

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Effect of myoelectric biofeedback therapy on upper limb function in elderly patients with cerebral infarction | Within 3 days of hospitalization, on the 1 day of discharge, one month after discharge
  Fugl-Meyer Functional Score (FMA) is evaluated, and the higher the score, the stronger the motor function.

SECONDARY OUTCOMES:
Influence on stroke quality of life in elderly patients with cerebral infarction | Within 3 days of hospitalization, on the 1 day of discharge, one month after discharge
  Assessment of Daily Living Ability Scale (ADL)is evaluated,The higher the score, the greater the independence of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yinkai Cheng, Study Chair — The Fourth Affiliated Hospital Zhejiang University School of Medicine
Locations (1):
- Yinkai Cheng, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No